CLINICAL TRIAL: NCT00005306
Title: Natural History of Post-transfusion Non-A, Non-B Hepatitis
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 3007
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2004-08

CONDITIONS: Hepatitis, Viral, Human; Blood Transfusion; Liver Diseases
MeSH Terms: conditions — Hepatitis, Viral, Human; Liver Diseases

SUMMARY:
To compare the clinical, biochemical, and histological status of Non-A, Non-B post-transfusion hepatitis patients with that of patients who did not develop post-transfusion hepatitis.

DETAILED DESCRIPTION:
BACKGROUND:

Hepatitis following the transfusion of blood and blood products continues to be an important problem, despite routine hepatitis surface antigen (HBsAg) screening of donor blood. In the mid 1980s, seven to ten percent of transfused individuals developed post-transfusion hepatitis (PTH). The majority of the cases were ascribed to the virus(es) of NANB hepatitis. Because the viral agent or agents responsible for this disease had not been identified in 1988, it was not possible to prevent the illness. There was evidence that the incidence of NANB PTH could be reduced by the use of volunteer donor blood instead of commercial blood. Other measures, in the absence of a specific test, related to efforts to develop a surrogate test to screen donor blood. The most promising approach in 1988 was to measure ALT activity and to exclude donors with increased levels of the enzyme. The measurement of antihepatitis-B core antigen (anti-HBc) was another surrogate test that appeared to be useful. Acute hepatitis caused by this agent(s) is mild and often asymptomatic, although in rare instances fulminant hepatitis may result and indeed may be associated with a higher mortality than that occurring in the course of acute hepatitis A or B.

Of greater concern was the finding that chronic hepatitis appeared to be a common outcome of acute NANB PTH. Chronic NANB hepatitis was defined as the presence of chronic liver disease in a patient who was negative for the serologic markers of hepatitis B virus, hepatitis A virus, cytomegalovirus, and Epstein-Barr virus, and who did not have a history of drug toxicity, alcoholism, or heart failure.

It appeared likely that chronic liver disease occurred at least as commonly, and perhaps more commonly, following infection with the NANB virus(es) than with the hepatitis B virus. Furthermore, evidence suggested that the presumed serious histopathologic abnormalities of chronic active hepatitis and cirrhosis were also more common.

The chronic sequelae of NANB hepatitis infection may therefore be more important than the acute illness. That information was of profound importance to blood bankers. Because the most disturbing data had been derived primarily from isolated studies, suggesting possible regional overtones or an effect of large volume transfusion, it seemed appropriate to study the problem of chronic NANB hepatitis on a wider scale.

DESIGN NARRATIVE:

The design was that of a retrospective, prospective study which followed two previously studied cohorts. In Phase I, evidence was presented that subjects in the Transfusion-Transmitted Virus Study and the Veterans Administration Cooperative Study of Post-transfusion Hepatitis could be located and their current status established. Initiation of Phase II was dependent on successful completion of Phase I.

In Phase II, medical records of all individuals identified in Phase I were obtained. The records were examined for clinical morbidity and mortality with particular attention given to liver-related abnormalities. Death certificates were sought for deceased patients. All surviving patients in the control and case groups were invited to participate and were re-evaluated and followed prospectively. Controls were matched for age, race, gender, and number of units of blood product received. Initial re-evaluation consisted of a medical history, physical examination, and a series of biochemical tests for evidence of chronic liver disease. In the initial evaluation, survivors were compared for clinical evidence of chronic liver disease, biochemical, and special test evidence of chronic liver disease.

In Phase III, all subjects from both groups were followed for six months by biochemical screening, including aminotransferase (ALT) and aspartate aminotransferase (AST). Enzyme assays were performed at least three times, thirty days apart. If aminotransferase activity was persistently abnormal, a liver biopsy was performed. The initial six month follow-up was designed to detect chronic liver disease. Once evidence of chronic liver disease had been established, those patients with chronic liver disease and controls were re-evaluated for evidence of liver disease at six-month intervals for three years from the initial visit.

The study was renewed in 1993 in order to develop a protocol and manual of operations for continuation of the study on the long- term follow-up of transfusion-associated non-A,non-B (NANB) hepatitis; to conduct annual National Death Index (NDI) searches for all cohort members who were alive or not located at last follow-up; to obtain and code death certificates for all newly deceased; and to collect and abstract medical records for all hospitalizations that occurred since the last follow-up for newly deceased subjects. The searches were conducted to determine whether a mortality difference between the infected cohort and the controls would develop with longer observation, as was suggested by the continued presence of chronic liver disease. Each surviving member was contacted annually, and medical records for all hospitalizations that occurred since the last follow-up for those subjects who reported liver disease were collected and abstracted. The contacts ensured that any liver disease that may have been missed through enzyme screening, or which may have newly developed, would be identified.

The study was formerly supported by N01HB87047.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1988-03; Study Completion 2001-09

CONTACTS AND LOCATIONS:
Overall Officials: Leonard Seeff — Georgetown University

REFERENCES:
- [Background] Seeff LB, Buskell-Bales Z, Wright EC, Durako SJ, Alter HJ, Iber FL, Hollinger FB, Gitnick G, Knodell RG, Perrillo RP, et al. Long-term mortality after transfusion-associated non-A, non-B hepatitis. The National Heart, Lung, and Blood Institute Study Group. N Engl J Med. 1992 Dec 31;327(27):1906-11. doi: 10.1056/NEJM199212313272703. PMID 1454085
- [Background] Duffy LF, Kerzner B, Seeff L, Barr SB, Soldin SJ. Preliminary assessment of glycine conjugation of para-aminobenzoic acid as a quantitative test of liver function. Clin Biochem. 1995 Oct;28(5):527-30. doi: 10.1016/0009-9120(95)00036-9. PMID 8582052
- [Background] Koff RS, Seeff LB. Economic modeling of treatment in chronic hepatitis B and chronic hepatitis C: promises and limitations. Hepatology. 1995 Dec;22(6):1880-2. No abstract available. PMID 7490001
- [Background] Tedeschi V, Seeff LB. Diagnostic tests for hepatitis C: where are we now? Ann Intern Med. 1995 Sep 1;123(5):383-5. doi: 10.7326/0003-4819-123-5-199509010-00009. No abstract available. PMID 7625627
- [Background] Seeff LB. Natural history of viral hepatitis, type C. Semin Gastrointest Dis. 1995 Jan;6(1):20-7. No abstract available. PMID 7894963
- [Background] Seeff LB, Alter HJ. Spousal transmission of the hepatitis C virus? Ann Intern Med. 1994 May 1;120(9):807-9. doi: 10.7326/0003-4819-120-9-199405010-00014. No abstract available. PMID 8147555
- [Background] Norman JE, Beebe GW, Hoofnagle JH, Seeff LB. Mortality follow-up of the 1942 epidemic of hepatitis B in the U.S. Army. Hepatology. 1993 Oct;18(4):790-7. doi: 10.1002/hep.1840180407. PMID 8406352
- [Background] Seeff LB, Hollinger FB, Alter HJ, Wright EC, Cain CM, Buskell ZJ, Ishak KG, Iber FL, Toro D, Samanta A, Koretz RL, Perrillo RP, Goodman ZD, Knodell RG, Gitnick G, Morgan TR, Schiff ER, Lasky S, Stevens C, Vlahcevic RZ, Weinshel E, Tanwandee T, Lin HJ, Barbosa L. Long-term mortality and morbidity of transfusion-associated non-A, non-B, and type C hepatitis: A National Heart, Lung, and Blood Institute collaborative study. Hepatology. 2001 Feb;33(2):455-63. doi: 10.1053/jhep.2001.21905. PMID 11172349
- [Background] Lin HJ, Seeff LB, Barbosa L, Hollinger FB. Occurrence of identical hypervariable region 1 sequences of hepatitis C virus in transfusion recipients and their respective blood donors: divergence over time. Hepatology. 2001 Aug;34(2):424-9. doi: 10.1053/jhep.2001.26635. PMID 11481629
- [Background] Harris DR, Gonin R, Alter HJ, Wright EC, Buskell ZJ, Hollinger FB, Seeff LB; National Heart, Lung, and Blood Institute Study Group. The relationship of acute transfusion-associated hepatitis to the development of cirrhosis in the presence of alcohol abuse. Ann Intern Med. 2001 Jan 16;134(2):120-4. doi: 10.7326/0003-4819-134-2-200101160-00012. PMID 11177315
- Available data/document: Individual Participant Data Set: NANB-TAH — http://biolincc.nhlbi.nih.gov/studies/NANB-TAH/ — NHLBI provides controlled access to IPD through BioLINCC. Access requires registration, evidence of local IRB approval or certification of exemption from IRB review, and completion of a data use agreement.
- Available data/document: Study Forms — http://biolincc.nhlbi.nih.gov/studies/NANB-TAH/